CLINICAL TRIAL: NCT05109637
Title: Study to Assess the Clinical Validity of Konectom™ in Adults Living With Neuromuscular Disorders
Brief Title: A Study to Assess the Clinical Validity of Konectom™ in Adults Living With Neuromuscular Disorders
Acronym: DigiNOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DE-SMG-11894; CIV-21-06-036845 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Neuromuscular Diseases; Spinal Muscular Atrophy; Digital technology; Digital outcome assessments; Smartphone; Digital Biomarkers
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with SMA (PwSMA) (Experimental): Participants with SMA will have their motor functions assessed using the Konectom NMD smartphone-based application up to Day 28.
  Interventions: Device: Konectom NMD Application
- Participants with ALS (PwALS) (Experimental): Participants with ALS will have their cognitive and motor functions assessed using the Konectom NMD smartphone-based application up to Day 28.
  As per protocol version 4.0, enrolment of ALS participants is stopped, and the data of the already enrolled ALS participants would not be analyzed.
  Interventions: Device: Konectom NMD Application
- Healthy Participants (Experimental): Healthy participants will have their cognitive and motor functions assessed using the Konectom NMD smartphone-based application for 28 days.
  Interventions: Device: Konectom NMD Application

INTERVENTIONS:
Device: Konectom NMD Application — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to explore the convergent validity of smartphone-based Konectom DOAs against in-clinic standard assessments.

The secondary objectives of this study are to evaluate the test-retest reliability of smartphone-based Konectom Digital Outcome Assessments (DOAs); to determine the relationship between Konectom upper limb DOAs and conventional upper limb assessments in clinical environments; to determine the relationship between Konectom lower limb DOAs and status of ambulation in clinical environments; to evaluate group differences in smartphone-based Konectom DOAs [self-administered at home and in-clinic] between person with spinal muscular atrophy (PwSMA) and healthy subjects (HS); to evaluate the variability of Konectom DOAs self-administered in everyday environment in HS and PwSMA; to compare Konectom DOAs between in-clinic supervised administration versus self-assessments in everyday environment in HS, PwSMA groups; to evaluate the relationship of Konectom DOAs against patient-reported outcomes (PROs) in PwSMA and to evaluate the clinical safety of Konectom in PwSMA.

ELIGIBILITY:
Key Inclusion Criteria:

For PwSMA

* Genetic documentation of 5q SMA (homozygous gene deletion, mutation, or compound heterozygote).

For Healthy Participants

* Age group matched with SMA participants

Key Exclusion Criteria:

For PwSMA

* Change of disease modifying treatment (DMT) in the last 1 month.
* Recent history of bacterial meningitis, viral encephalitis, or hydrocephalus.
* Addiction (alcohol or another drug abuse).
* Presence of an implanted shunt for the drainage of cerebrospinal fluid (CSF) or of an implanted central nervous system (CNS) catheter.
* Hospitalization for surgery (i.e., scoliosis surgery or other surgery), pulmonary event, or nutritional support in the previous 2 months or planned within the study duration.
* Known pregnancy.

NOTE: Other protocol defined inclusion/ exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Type of Correlation of Konectom DOAs Versus Hammersmith Functional Motor Scale-Expanded (HFMSE) Total Score in PwSMA | Up to 28 days
  This outcome measure will assess the convergent validity of smartphone-based Konectom DOAs against in-clinic standard assessments.
Strength of Correlation of Konectom DOAs Versus HFMSE Total Score in PwSMA | Up to 28 days
  This outcome measure will assess the convergent validity of smartphone-based Konectom DOAs against in-clinic standard assessments.

SECONDARY OUTCOMES:
Interclass Correlation Coefficient (ICC) of the Konectom Digital Outcome Assessment (DOA) Scores | Up to 28 days
  This outcome measure will assess test-retest reliability of smartphone-based Konectom DOAs.
Type of Correlation of Upper Limb Konectom DOAs Versus Revised Upper Limb Module (RULM) in PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Upper Limb DOAs and conventional upper limb assessments in clinical environments.
Strength of Correlation of Upper Limb Konectom DOAs Versus RULM in PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Upper Limb DOAs and conventional upper limb assessments in clinical environments.
Type of Correlation of Upper Limb Konectom DOAs Versus 9-Hole Peg test (9HPT) in PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Upper Limb DOAs and conventional upper limb assessments in clinical environments.
Strength of Correlation of Upper Limb Konectom DOAs Versus 9HPT in PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Upper Limb DOAs and conventional upper limb assessments in clinical environments.
Type of Correlation of Lower Limb Konectom DOAs Versus 6-Minute Walk Test (MWT) Total Distance in Ambulatory PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Lower Limb DOAs and status of ambulation in clinical environments.
Strength of Correlation of Lower Limb Konectom DOAs Versus 6-MWT Total Distance in Ambulatory PwSMA | Up to 28 days
  This outcome measure will assess the relationship between Konectom Lower Limb DOAs and status of ambulation in clinical environments.
Differences Between PwSMA and HS in the Konectom DOA Scores During Each Testing Condition | Up to 28 days
  This outcome measure will assess the group differences in smartphone-based Konectom DOAs [self-administered at home and in-clinic] between PwSMA and healthy subjects (HS).
Standard Deviation of Each Participant's Raw Konectom DOA Scores Over the At-Home Period | Up to 28 days
  This outcome measure will assess the variability of Konectom DOAs self-administered in everyday environment in HS and PwSMA.
Paired-Comparisons of Konectom DOA Scores Between In-Clinic Supervised Administration and Self-Assessment In Everyday Environment, Separately for HS and PwSMA Groups | Up to 28 days
  This outcome measure will assess the comparison of Konectom DOAs between in-clinic supervised administration versus self-assessments in everyday environment in HS and PwSMA groups.
Type of Correlation of Konectom DOA Scores Versus Neuro-Quality of Life (QoL) Total Scores in PwSMA | Up to 28 days
  This outcome measure will assess the relationship of Konectom DOAs against patient-reported outcomes (PROs) in PwSMA.
Strength of Correlation of Konectom DOA Scores Versus Neuro-QoL Total Scores in PwSMA | Up to 28 days
  This outcome measure will assess the relationship of Konectom DOAs against PROs in PwSMA.
Type of Correlation of Konectom DOA Scores Versus Fatigue Severity Scale (FSS) Total Scores in PwSMA | Up to 28 days
  This outcome measure will assess the relationship of Konectom DOAs against PROs in PwSMA.
Strength of Correlation of Konectom DOA Scores Versus FSS Total Scores in PwSMA | Up to 28 days
  This outcome measure will assess the relationship of Konectom DOAs against PROs in PwSMA.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) Related to Konectom NMD Use | Up to 43 days
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the Investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect. This outcome measure will assess the clinical safety of Konectom NMD in PwSMA.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- Germany (5):
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Dresden
  - Research Site, Hanover
  - Research Site, Heidelberg
  - LMU Klinikum Friedrich-Baur-Institute, Dept. of Neurology, Munich

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/